CLINICAL TRIAL: NCT06530810
Title: A Phase 1b, Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10382 Combination Therapy in Patients With Chronic Myeloid Leukemia
Brief Title: Study of HS-10382 Combination in Patients With Chronic Myeloid Leukemia (CML)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10382-102
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Chronic Myelogenous Leukemia; CML Chronic Phase; CML Accelerated Phase
Keywords: CML-CP/AP; HS-10382; Flumatinib; Allosteric inhibitor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10382+Flumatinib (Experimental): Subjects with resistant or intolerant CML CP/AP will be enrolled in dose-escalation stage.Dose escalation of HS-10382 combined flumatinib will be done to determine maximum tolerated dose(Part 1).
  Depending on data obtained from the dose-escalation stage,dose expansion may proceed with in subjects with newly diagnosed CML-CP.The safety and efficacy will be evaluated at the target dose.(Part 2)
  Interventions: Drug: HS-10382+Flumatinib

INTERVENTIONS:
Drug: HS-10382+Flumatinib — Drug:HS-10382+Flumatinib HS-10382 is administered orally BID Drug:Flumatinib Flumatinib 400mg once daily

SUMMARY:
HS-10382 is a small molecular, oral potent, allosteric inhibitor. By binding a myristoyl site of the BCR-ABL1 protein, HS-10382 locks BCR-ABL1 into an inactive conformation. Flumatinib is the first approved second generation TKI in China and a derivative of imatinib.

The primary objective of this study is to evaluation the safety and tolerability and of HS-10382 combination therapy in patients with chronic myeloid leukemia (CML).

The secondary objectives is to evaluate the PK profile, major metabolites and efficacy of HS-10382 in CML-CP/AP subjects after combination therapy, and to explore the kinase domain mutations associated with TKI resistance

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Men or women aged more than or equal to (≥) 18 years, and less than (<) 75 years.
* CML-CP/AP patients with the Ph chromosome or BCR-ABL1 fusion genes.
* Patient with CML-CP/AP who are resistant to or intolerant to previous TKIs therapy.
* ECOG performance status of 0-1 and no worsening within 2 weeks before the first dose.
* Life expectancy ≥ 12 weeks.
* Men or women should be using adequate contraceptive measures throughout the study; Females should not be breastfeeding at the time of screening, during the study and until 6 months after completion of the study.
* Females must have evidence of non-childbearing potential.

Exclusion Criteria:

* CML-CP patients who have acquired CCyR and have not lost it.
* Patients with CML-CP who have progressed to AP or blast phase(BP.)
* Patients with CML-AP who have obtained CHR or no evidence of CML in peripheral blood.
* Patients with CML-AP who have progressed to BP.
* Previous treatment with a BCR-ABL1 TKI allosteric inhibitor .
* Impaired cardiac function including any one of the following:
* Resting corrected QT interval (QTc) > 470 ms obtained from electrocardiogram (ECG), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG.
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events,
* Left ventricular ejection fraction (LVEF) ≤ 50%.
* Myocardial infarction occurred within 6 months of the first scheduled dose of study drug.;
* Congestive heart failure occurred within 6 months of the first scheduled dose of study drug.;
* Uncontrollable angina.
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* Any severe or uncontrolled systemic diseases (i.e. uncontrolled hypertension or diabetes).
* Clinically severe gastrointestinal dysfunction that may affect drug intake, transport or absorption.
* Severe infection within 4 weeks prior to the first scheduled dose of study drug
* Inadequate other organ function.
* History of other malignancies.
* History of hypersensitivity to any active or inactive ingredient of HS-10382 and flumatinib.
* History of neuropathy or mental disorders, including epilepsy and dementia.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for HS-10382 combined treatment | Up to day 28 from the first dose
  MTD was defined as the previous dose level at which 2 out of 3 subjects or 2 out of 6 subjects experienced a DLT

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Cycle 1 day 1 up to 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0
maximum plasma concentration of HS-10382 or Flumatinib(and its major metabolite ) after HS-10382 combination therapy | Cycle 1 day 1 up to 28 days after the last dose
  Cmax is the maximum observed concentration.
Time to reach maximum plasma concentration of HS-10382 or Flumatinib(and its major metabolite) after HS-10382 combination therapy | Cycle 1 day 1 up to 28 days after the last dose
  Tmax is defined as time to reach maximum observed plasma concentration
half-life (T1/2) of HS-10382 combination therapy | Cycle 1 day 1 up to 28 days after the last dose
  half-life is the time measured for the concentration to decrease by one half
Area under the curve (AUC) of HS-10382 combination therapy | Cycle 1 day 1 up to 28 days after the last dose
  The AUC is defined as the area under the plasma concentration-time curve
Hematologic Response of combination therapy with HS-10382 | up to 24 months
  To record and analyse the hematologic response of subjects. Hematologic response will be assessed by complete blood count (CBC) and physical examination at each visit.
Cytogenetic Response of combination therapy with HS-10382 | up to 24 months
  To record and analyse the cytogenetic response of subjects. Cytogenetic response (CyR) is based on the prevalence of Ph+ cells in metaphase from bone marrow (BM) sample.
Molecular Response of combination therapy with HS-10382 | up to 24 months
  To record and analyse the molecular response of subjects. Molecular response will be assessed by BCR-ABL1 transcript level as measured by RQ-PCR.
Event-free survival (EFS) | up to 24 months
  EFS is defined as the time from the date of first dose to the earliest occurrence of the following events: death due to any cause ; loss of CHR ,loss of PCyR ;loss of CCyR ; discontinuation of study treatment due to AE or treatment failure ; progression to AP/BC .
Progression-free survival (PFS) | From the first dose to disease progression or withdrawal from study, whichever came first,up to 24 months
  PFS is defined as the time from the date of first dose to the earliest occurrence of progression to AP/BC or death from any cause.
Overall survival (OS) | From the first dose up to death or withdrawal from study, whichever came first, up to 24 months
  OS is defined as the time from the date of first dose to the date of death from any cause.

IPD SHARING:
Plan to Share IPD: No